CLINICAL TRIAL: NCT03437109
Title: Clinical and Epidemiological Characteristics and Efficacy of Androgen Substitution for Hypogonadism in Men With Type 2 Diabetes Mellitus Under Routine Clinical Practice
Brief Title: Efficacy of Androgen Substitution for Hypogonadism in Men With Type 2 Diabetes Mellitus
Acronym: DESTINY
Status: Completed | Type: Observational
Sponsor: Besins Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: BH-DM-11-2017
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Hypogonadism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laboratory tests — Testosterone HSBG Hb1Ac LH

SUMMARY:
The purpose of the study is to get data of prevalence of testosterone deficiency in patient with T2DM in Russian Federation

DETAILED DESCRIPTION:
Clinical and Epidemiological Characteristics and Efficacy of Androgen Substitution for Hypogonadism in Men With Type 2 Diabetes Mellitus Under Routine Clinical Practice (DESTINY)

ELIGIBILITY:
Inclusion Criteria:

* Male 45-60 years old
* Diagnosis of T2DM according to approved standards
* Signed Informed Consent Form

Exclusion Criteria:

* Prepubertal hypogonadism of any genesis;
* Sexual and developmental disorders;
* Absence of at least one of the testicles;
* Cryptorchidism, including in the anamnesis;
* Injuries and / or surgical interventions on the genitals with loss of at least one of the testicles;
* Established diagnosis of panhypopituitarism in accordance with current recommendations / standards;
* Androgen therapy, administered at the time of the study or in the anamnesis;
* Admission of anabolic steroids;
* Alcoholism or drug addiction;
* Insolvency.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men with T2DM aged between 45-60 years old
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of hypogonadism in patients with T2DM | 2017-2018
  The prevalence of hypogonadism in patients with T2DM

CONTACTS AND LOCATIONS:
Overall Officials: Marina SHESTAKOVA, academitian, Study Chair — ENC
Locations (2):
- Russia (2):
  - ENC, Moscow
  - Central Clinical Hospital, Moscow

IPD SHARING:
Plan to Share IPD: Undecided